CLINICAL TRIAL: NCT06938932
Title: Exposure to Environmental Heat and Intervention Study
Brief Title: Effects of Environmental Heat Exposure on Human Multiple Organ Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yinan Qu (Other)
Collaborators: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor-Investigator, Yinan Qu, Master, Shandong University
Organization: Shandong University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: LL20241102
Record Dates: First submitted 2025-04-04; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Heat Stress Disorders; Wounds and Injuries; Body Temperature Changes; Multiple Organ Dysfunction
MeSH Terms: conditions — Heat Stress Disorders; Wounds and Injuries; Body Temperature Changes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be informed of the study interventions before providing informed consent but will be masked to the order of exposure (i.e., participants will not know the exposure conditions). Data will be blinded prior to analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High temperature group (Experimental): This group including 24 healthy subjects will be exposed to high temperature for about 3 hours in a chamber.
  Interventions: Other: High temperature exposure
- Moderate temperature group (Sham Comparator): This group including 24 healthy subjects will be exposed to moderate temperature for about 3 hours in a chamber.
  Interventions: Other: Moderate temperature exposure

INTERVENTIONS:
Other: High temperature exposure — Subjects will be exposed to 35 degree Celsius and 45% relative humidity for 3 hours, resting during the whole periods.
  Arms: High temperature group
Other: Moderate temperature exposure — Subjects will be exposed to 24degree Celsius and 45% relative humidity for 3 hours, resting during the whole periods.
  Arms: Moderate temperature group

SUMMARY:
This is a randomized controlled human exposure crossover study. Investigators aims to assess the acute effects of high temperature exposure and the underlying mechanisms.

DETAILED DESCRIPTION:
The objective of this study is to study changes in functions of multiple organs under heat exposure, which mainly include changes of cardiac function and lung function. In addition, biological samples such as blood samples, nasal fluid, and urine, etc were collected to explore changes in biomarkers such as complete blood count, liver function, kidney function, and inflammatory indicators, etc. Biochemical analysis and omics analysis were conducted to study the changes of human physiological function caused by heat exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese nationality（aged 18-30 years healthy males and females）;
2. With ability to read and understand Chinese smoothly;
3. Living in Jinan during the study period;
4. Body mass index ≥ 18.5 and ≤ 28;
5. Normal resting ECG；
6. Normal lung function: i. Forced vital capacity (FVC)≥80% of that predicted for gender, ethnicity, age and height; ii. Forced expiratory volume in one second (FEV1) ≥80% of that predicted for gender, ethnicity, age and height; iii. FEV1/FVC ratio≥80% of predicted values.

Exclusion Criteria:

1. Medications or dietary supplements intake that may alter body temperature during the study period;
2. Individuals who have unspecified illnesses, which in the judgment of the investigators might increase the risk associated with heat exposure will be a basis for exclusion;
3. Subjects with anemia, needle fainting and other signs unsuitable for blood drawing；
4. Subjects with cardiovascular diseases or other chronic medical condition, such as congenital heart disease, pulmonary heart disease, and hypertension, etc;
5. Subjects with a history of major cardio-vascular, respiratory, or nervous system surgery, etc;
6. Subjects with neurologic disorders, such as stroke, traumatic brain injury, epilepsy, and depression;
7. Subjects with allergic diseases, such as allergic rhinitis and allergic asthma, etc;
8. Subjects are pregnant, attempting to become pregnant or breastfeeding;
9. Subjects who are currently smoking (including vaping, hookah and e-cigarette) or have smoking history within 1 year of study (defined as more than 1 pk/yr in the past year) or have a greater than equal to a 5 pack year smoking history;
10. Subjects living with a smoker who smokes inside the house;
11. Subjects who are current drinking or have frequent alcohol use (defined as at least 1 time per week) in the past 6 months;
12. Provisional exclusion criteria, such as acute infection in the past two weeks or taking antibiotics. (Subjects can be enrolled after 2 weeks)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-21 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure | Systolic and diastolic blood pressure will be measured within 15 minutes before exposure and immediately after the exposure session, and every 15 minutes during exposure.
  Brachial arterial blood pressure will be measured
Cardiac output | Cardiac output will be checked within half an hour before exposure and immediately after exposure.
  Cardiac output will be measured by heart color ultrasound
Heart rate variability | Cardiac variability will be monitored in real time from half an hour before exposure to half an hour after exposure, with data automatically recorded every 8 seconds.
  Heart rate variability will be measured using 24-hour holter electrocardiogram
Change of forced expired volume in the first second (FEV1) | FEV1 will be checked within half an hour before exposure and 15 minutes after exposure.
  The changes of FEV1 will be measured by a smart spirometer. Before the pulmonary function test, subjects will practice several times by themselves. During the examination, each subject stands and clamps the nose clip, and repeats the test, with the best result as the criterion.
Changes of forced vital capacity (FVC) | FVC will be checked within half an hour before exposure and 15 minutes after exposure.
  The changes of FVC will be measured by a smart spirometer.
Changes of peak expiratory flow rate (PEF) | PEF will be checked within half an hour before exposure and 15 minutes after exposure.
  The changes of PEF will be measured by a smart spirometer.
Changes of maximum expiratory flow rate at 25% vital capacity (MEF25) | MEF25 will be checked within half an hour before exposure and 15 minutes after exposure.
  The changes of MEF25 will be measured by a smart spirometer.
Changes of maximum expiratory flow rate at 50% vital capacity (MEF50) | MEF50 will be checked within half an hour before exposure and 15 minutes after exposure.
  The changes of MEF50 will be measured by a smart spirometer.
Changes of maximum expiratory flow rate at 75% vital capacity (MEF75) | MEF75 will be checked within half an hour before exposure and 15 minutes after exposure.
  The changes of MEF75 will be measured by a smart spirometer.

SECONDARY OUTCOMES:
Differences in metabolic profiling detected in blood between the two exposures and before and after each exposure | Prior to and 1 hour after exposure
  The differential metabolic profiling in peripheral blood related to high temperature exposure will be detected by mass spectrometry-based non-targeted metabolomics.
Differences in transcriptome detected in blood between the two exposures and before and after each exposure | Prior to and 1 hour after exposure
  The differential transcriptome in peripheral blood related to high temperature exposure will be detected by mass spectrometry-based non-targeted transcriptomics.
Differences in proteome detected in blood between the two exposures and before and after each exposure | Prior to and 1 hour after exposure
  The differentially expressed proteins in peripheral blood related to high temperature exposure will be detected by non-targeted proteomics
EEG power in α band | EEG power in α band will be measured immediately during the same exposure period the day before exposure and within half an hour of the end of the exposure day.
  EEG power in α band will be monitored by EEG measuring instrument
EEG power in θ band | EEG power in θ band will be measured immediately during the same exposure period the day before exposure and within half an hour of the end of the exposure day.
  EEG power in θ band will be monitored by EEG measuring instrument
EEG power in β band | EEG power in β band will be measured immediately during the same exposure period the day before exposure and within half an hour of the end of the exposure day.
  EEG power in β band will be monitored by EEG measuring instrument
EEG power in δ band | EEG power in δ band will be measured immediately during the same exposure period the day before exposure and within half an hour of the end of the exposure day.
  EEG power in δ band will be monitored by EEG measuring instrument
Response event-related potentials (ERPs) | ERPs will be measured immediately during the same exposure period the day before exposure and within half an hour of the end of the exposure day.
  ERPs will be monitored by EEG measuring instrument, including P300, N1/P1 and so on.
Frequency domain and energy ratio index, θ/β ratio | θ/β ratio will be measured immediately during the same exposure period the day before exposure and within half an hour of the end of the exposure day.
  θ/β ratio will be monitored by EEG measuring instrument, which is an important parameter for response frequency domain and energy ratio index
Cerebral blood flow changes | Cerebral blood flow changes will be examed within half an hour before exposure and half an hour after exposure.
  Cerebral blood flow changes will be measured by transcranial doppler

OTHER OUTCOMES:
Change in tumor necrosis factor-α (TNF-α) concentrations | Prior to and 1 hour after exposure
  TNF-α will be tested through blood samples
Change in C reactive protein (CRP) concentrations | Prior to and 1 hour after exposure
  CRP will be tested through blood samples
Change in interleukin-6 (IL-6) concentrations | Prior to and 1 hour after exposure
  IL-6 will be tested through blood samples
Change in interleukin-1β (IL-1β) concentrations | Prior to and 1 hour after exposure
  IL-1β will be tested through blood samples
Change in liver function indicators | Prior to and 1 hour after exposure
  Liver function indexes will be tested through blood samples, including glutamic-pyruvic transaminase (ALT), glutamic oxalacetic transaminase (AST), glutamyltranspeptidase (GGT), alkaline phosphatase (ALP), total protein (TP), albumin(ALB), total bilirubin (TBIL), direct bilirubin (DBIL) and so on.
Change in kidney function indicators | Prior to and 1 hour after exposure
  Liver function indexes will be tested through blood samples, including urea nitrogen (BUN), creatinine (CR), Cystatin C (CYS C) and so on.
Change in Uric Acid (UA) | Prior to and 1 hour after exposure
  UA will be tested through blood samples
Change in myocardial and vascular injury indicators | Prior to and 1 hour after exposure
  myocardial and vascular injury indicators will be tested through blood samples, including creatine kinase (CK), Creatine Kinase Isoenzyme (CKMB), lactic dehydrogenase (LDH), α-hydroxybutyrate kinase and so on.
Change in coagulation indicators | Prior to and 1 hour after exposure
  Coagulation indicators will be tested through prothrombin time(PT), activated partial thromboplastin time (APTT), plasma fibrinogen (FIB), thrombin time (TT) and so on.
Blood routine examination | Prior to and 1 hour after exposure
  A routine test in the blood test, including red blood cells, white blood cells, platelets and other aspects of the test.
Routine urianlysis | Prior to and 1 hour after exposure
  A routine test in the urine sample, including urine specific gravity and so on.
Change in D-lactic acid | Prior to and 1 hour after exposure
  D-lactic acid will be tested through blood samples
Change in diamine oxidase(DAO) | Prior to and 1 hour after exposure
  DAO will be tested through blood samples
Weight | Prior to exposure and immediately after the exposure session
  Weight will be measured using a scale, wearing only short-sleeved shorts and slippers

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No